CLINICAL TRIAL: NCT04923594
Title: A Four-week, Double-blind, Placebo-controlled, Randomized, Multicenter, Parallel-group Study of the Safety and Efficacy of NLS-2 (Mazindol Extended Release) in Adults for the Treatment of Narcolepsy
Brief Title: Four-week Study of the Safety and Efficacy of NLS-2 (Mazindol Extended Release) in the Treatment of Narcolepsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NLS Pharmaceutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NLS-1021
Record Dates: First submitted 2021-06-09; First posted 2021-06-11 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Narcolepsy; Excessive Daytime Sleepiness; Cataplexy Narcolepsy
MeSH Terms: conditions — Narcolepsy; Disorders of Excessive Somnolence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NLS-2 (mazindol extended release) (Active Comparator): 2 mg dosed orally, once daily for 1 week; followed by 3 mg dosed orally, once daily for up to 3 weeks (total of 4 weeks)
  Interventions: Drug: mazindol extended release
- Placebo (Placebo Comparator): Dosed orally, once daily for up to 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: mazindol extended release — Dosed orally, once daily for up to 3 weeks
  Other Names: NLS-2
  Arms: NLS-2 (mazindol extended release)
Drug: Placebo — Dosed orally, once daily for up to 4 weeks.
  Arms: Placebo

SUMMARY:
This is a double-blind, randomized, placebo-controlled, multicenter trial of NLS-2 in adult patients with narcolepsy. The study will enroll approximately 60 patients and eligible patients will be treated to receive either NLS-2 or placebo for 4-weeks.

ELIGIBILITY:
Key Inclusion Criteria:

* Males and females between 18 and 65 years of age, inclusive
* Diagnosis of narcolepsy according to ICSD-3 (International Classification of Sleep Disorders, 3rd Edition) or Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria
* Body mass index from 18 to 40 kg/m2, inclusive
* Consent to use a medically acceptable method of contraception
* Willing and able to provide written informed consent

Key Exclusion Criteria:

* Female subjects who are pregnant, nursing, or lactating
* Any other clinically relevant medical, behavioral, or psychiatric disorder other than narcolepsy that is associated with excessive sleepiness
* History or presence of bipolar disorder, bipolar related disorders, schizophrenia, schizophrenia spectrum disorders, or other psychotic disorders according to DSM-5 criteria
* Use of any over-the-counter (OTC) or prescription medications that could affect the evaluation of excessive sleepiness
* Use of any medications that could affect the evaluation of cataplexy
* Received an investigational drug in the past 30 days or five half-lives (whichever is longer)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change in ESS Score From Baseline to Week 4 | Baseline to Week 4
  Change in Epworth Sleepiness Scale (ESS) score from Baseline to Week 4. A negative change from baseline represents improvement in excessive sleepiness.
  The ESS is a self-administered questionnaire with 8 questions. Each activity is scored on a scale ranging from 0-3, with 0 = would never fall asleep, and 3 = high chance of falling asleep. The total score ranges from 0-24, with a higher number representing an increased propensity for sleepiness.

SECONDARY OUTCOMES:
Subjects Reported Improved on the Patient Global Impression of Change (PGIc) at Week 4 | Baseline to Week 4
  Percentage of subjects reported as improved (minimally, much, or very much) on the PGIc at Week 4. PGIc is rated by subjects and measures the change in their condition since treatment starts on a 7-point scale ranging from 1= very much improved to 7= very much worse

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Camozzi, MD, Study Director — NLS Pharmaceutics
Locations (22):
- United States (22):
  - Sleep Disorders Center of Alabama, Birmingham, Alabama
  - Stanford Sleep Medicine Center, Redwood City, California
  - Pacific Research Network, San Diego, California
  - St. Francis Sleep Allergy and Lung Institute, Clearwater, Florida
  - Sleep Medicine Specialists of South Florida, Miami, Florida
  - Ivetmar Medical Group, Miami, Florida
  - The Angel Medical Research Corporation, Miami Lakes, Florida
  - Treken Primary care, Atlanta, Georgia
  - NeuroTrials Research, Atlanta, Georgia
  - Clinical Research Institute, Stockbridge, Georgia
  - Hawaii Pacific Neuroscience Clinical Research Center, Honolulu, Hawaii
  - The Center For Sleep & Wake Disorders, Chevy Chase, Maryland
  - Sleep and Attention Disorders, Sterling Heights, Michigan
  - Neurology and Sleep Disorders Clinic, Columbia, Missouri
  - Carolinas Sleep Specialists, Concord, North Carolina
  - Superior Clinical Research, LLC, Goldsboro, North Carolina
  - Advanced Respiratory and Sleep Medicine, Huntersville, North Carolina
  - Intrepid Research, Cincinnati, Ohio
  - Ohio Sleep Medicine Institute, Dublin, Ohio
  - Bogan Sleep Consultants, Columbia, South Carolina
  - Dharma PA d/b/a Southwest Family Medicine Associates, Dallas, Texas
  - Sleep Therapy & Research Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No